CLINICAL TRIAL: NCT02274844
Title: Improving Medication Adherence in the Alabama Black Belt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCORI-R-AD-1306-03565
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Coaching (Experimental): The intervention participants will receive the Living Well with Diabetes Program. The program will consist of educational DVDs with integrated storytelling about how community members accepted their disease and overcame barriers to medication adherence, plus one-on-one telephonic peer coaching.
  Interventions: Behavioral: Living Well with Diabetes Program
- Usual Care (No Intervention): At enrollment, the investigators will provide an educational DVD on general health and wellness topics including vaccination, cancer screening, osteoporosis and other topics not related to diabetes care. There will be no peer storytelling on these DVDs.

INTERVENTIONS:
Behavioral: Living Well with Diabetes Program — The intervention participants will receive the Living Well with Diabetes Program. The program will consist of educational DVDs with integrated storytelling about how community members accepted their disease and overcame barriers to medication adherence, plus one-on-one telephonic peer coaching
  Arms: Peer Coaching

SUMMARY:
Medication adherence is especially critical in regions like rural Alabama, where residents have among the worst health outcomes in the US. This project was designed in collaboration with our community member partners and builds on a 5-year partnership of community-engaged research on diabetes peer coaching interventions and our experience with peer storytelling. The investigators will test the hypothesis that an intervention designed within the Corbin and Strauss framework can improve adherence and health outcomes compared to usual care.

DETAILED DESCRIPTION:
Improving medication adherence is one of the greatest challenges in modern medicine. Despite decades of research on the topic, as many as half of patients with chronic diseases are not taking medications as recommended, and costs of nonadherence have been estimated at $290 billion annually. One reason for this persistent finding could be that interventions rarely acknowledge medications within the larger context of the lived experience of illness. Drawing on hundreds of patient interviews, Corbin and Strauss showed that chronic illness is a fundamentally destabilizing influence that forces us to confront the potential limitations of our "new", chronically ill self. Accepting our illness may be a crucial step in embracing medication adherence and other self-management behaviors as ways to restore balance following this disruption. The Corbin and Strauss framework is not often used to develop and test interventions to improve medication adherence, and this is the central objective of this proposal.

Medication adherence is especially critical in regions like rural Alabama, where residents have among the worst health outcomes in the US. Rates of cardiovascular mortality, diabetes and obesity are very high, but resources are scarce and the area's predominately black residents have deep-seated mistrust of the healthcare system (the region includes Tuskegee, site of the infamous syphilis study). This project was designed in collaboration with our community member partners and builds on a 5-year partnership of community-engaged research on diabetes peer coaching interventions and our experience with peer storytelling. The investigators will test the hypothesis that an intervention designed within the Corbin and Strauss framework can improve adherence and health outcomes compared to usual care. Our Aims are:

Aim 1: With our community partners, using qualitative research methods, build on already developed culturally tailored education material to develop the medication adherence intervention. The intervention will consist of educational DVDs with integrated storytelling about how community members accepted their disease and overcame barriers to medication adherence, plus one-on-one telephonic peer coaching. Activities include conducting focus groups with patients; creating the DVDs and the coaching intervention protocol; training peer coaches; and pilot testing.

Aim 2: Conduct a randomized controlled trial with 500 individuals with type 2 diabetes and medication nonadherence. The trial will compare the effect of usual care and the intervention on medication adherence and physiologic risk factors including A1c, blood pressure and low density lipoprotein cholesterol (primary outcomes), and quality of life and self-efficacy (secondary outcomes).

This innovative approach would be a major shift in how patients are helped in under resourced areas living with chronic diseases commit to taking medications, improving health and eventually reducing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* adults
* type 2 diabetes
* taking medications for diabetes
* medication non adherent

Exclusion Criteria:

* nursing home residence
* plans to move away in the next year
* advanced illnesses such as hemodialysis, cancer or dementia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika M Safford, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Univeristy of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data will stay at UAB

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment efforts in this area focused on attending health fairs, posting flyers at community locations such as libraries and churches. The main focus of recruitment was in the county's safety net clinic.
Period: Overall Study
Arm/Group | Peer Coaching | Usual Care
Started | 203 | 270
Completed | 165 | 238
Not Completed | 38 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Coaching | Usual Care | Total
Number analyzed (Participants) | 203 | 270 | 473
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.6) | 56.7 (12.1) | 57.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 212 | 371
  Male | 44 | 58 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 178 | 250 | 428
  All Others | 25 | 20 | 45
Marital Status [Count of Participants; unit: Participants] — Population: 1 subject in the usual care arm declined to provide this information.
  Participants
    number analyzed (Participants) | 203 | 269 | 472
    Married or living with partner | 75 | 94 | 169
    Never married, divorced, widowed, separated | 128 | 175 | 303
Annual Income [Count of Participants; unit: Participants] — Population: 10 subjects in the peer coaching arm and 11 subjects in the usual care arm declined to provide this information.
  Participants
    number analyzed (Participants) | 193 | 259 | 452
    <$20,000 | 133 | 185 | 318
    >=$20,000 | 60 | 74 | 134
Education [Count of Participants; unit: Participants] — Population: 1 subject in the peer coaching arm declined to provide this information.
  Participants
    number analyzed (Participants) | 202 | 270 | 472
    < High School | 46 | 51 | 97
    12th grade, GED, HS diploma | 69 | 99 | 168
    >High School | 87 | 120 | 207
Employment [Count of Participants; unit: Participants] — Population: 1 subject in the peer coaching arm and 2 subjects in the usual care arm declined to provide this information.
  Participants
    number analyzed (Participants) | 202 | 268 | 470
    Employed for wages or self-employed | 53 | 72 | 125
    Not worked(ret, out of wrk, homemker, unable work) | 149 | 196 | 345
HbA1c [Mean (Standard Deviation); unit: %] | 8.6 (2.2) | 8.3 (2.0) | 8.4 (2.1)
Hba1c [Count of Participants; unit: Participants]
  Less than 7.0 | 73 | 114 | 187
  7.0 or greater | 130 | 156 | 286
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 127.8 (19.4) | 129.1 (19.9) | 128.6 (19.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 36.4 (8.8) | 36.5 (8.0) | 36.5 (8.4)
Medication Adherence Score as measured by the Morisky Medication Adherence Scale [Count of Participants; unit: Participants] — 4-item Morisky Medication Adherence Scale-a validated assessment tool used to measure non-adherence. If subjects answered yes to 0 questions, this would indicate high adherence and if subjects answered yes to 4 questions, this would indicate low adherence.
  Participants
    Yes to 0 questions | 67 | 104 | 171
    Yes to 1 questions | 84 | 98 | 182
    Yes to 2 questions | 34 | 40 | 74
    Yes to 3 questions | 12 | 20 | 32
    Yes to 4 questions | 6 | 7 | 13
    Missing | 0 | 1 | 1
Number of Subjects Taking Insulin [Count of Participants; unit: Participants] | 96 | 111 | 207

OUTCOME MEASURES:

1. Primary Outcome: Change in Self Reported Medication Adherence
Description: Patient-reported adherence to medications as a medication adherence score, from 0-3, where a higher score indicates worse adherence.
Time Frame: Baseline, 6 months
Population: 39 participants in the peer coaching arm and 31 participants in the usual care arm were not analyzed because the participants were unable to be contacted, had health reasons, or did not have time.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 0.78 (0.80) | 0.74 (0.79)
  6 months | 0.53 (0.66) | 0.62 (0.76)
  Change at 6 months | -0.25 (0.70) | -0.12 (0.71)
Statistical Analysis 1: Comparison: Peer Coaching vs Usual Care; The study was powered to detect clinically meaningful differences in physiologic risk factors; it had four primary outcomes.Power estimates accounted for clustering of patients within towns, using a variance inflation factor, conservatively estimating power for ICC=0.01-0.05. Process measures were selected to understand which aspects of the intervention were particularly effective, assessing both program satisfaction and peer coach effectiveness; Test type: Superiority — The outcomes were all continuous or ordinal measures, thus unadjusted hypothesis tests used t-tests or the Wilcoxon-Mann-Whitney test, as appropriate, and statistical modeling used linear regression. ANCOVA was used to adjust for baseline covariates with imbalance across treatment arms (race) and baseline values of the measures; p = 0.22, ANCOVA — The main hypotheses tested were that intervention participants would have higher medication adherence and significantly greater improvement in A1c, BP, LDL-C, and measures of quality of life, and self-efficacy compared to control participants; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.23 to 0.05]

2. Primary Outcome: Change in Percentage of HbA1c
Description: Hemoglobin A1c test to identify the average amount of glucose (sugar) present in a patient's blood.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
percentage of HbA1c
  Baseline | 8.4 (2.11) | 8.3 (1.99)
  6 months | 8.1 (1.9) | 8.1 (1.8)
  Change at 6 months | -0.37 (1.71) | -0.24 (1.55)

3. Primary Outcome: Change in Blood Pressure
Description: 2 BP measures were taken 1 minute apart using a LifeSource UA-789 digital blood pressure monitor.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
mmHg
  Baseline | 128.5 (19.6) | 129.3 (19.5)
  6 months | 130.6 (20.7) | 133.6 (18.4)
  Change at 6 months | 2.5 (19.5) | 4.1 (20.5)

4. Primary Outcome: Change in Low-Density Lipoprotein (LDL) Cholesterol
Description: Finger stick, spectrophotometer to measure cholesterol level.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
mg/dL
  Baseline | 84.6 (38.4) | 80.7 (36.3)
  6 months | 80.1 (33.1) | 82.2 (31.0)
  Change at 6 months | -4.5 (38.6) | 1.5 (38.2)

5. Secondary Outcome: Change in Quality of Life as Assessed With the Short Form 12- Mental Component
Description: Short Form-12 Mental Component and Physical Component Summary scores range from 0-100; higher scores indicate greater quality of life.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 42.7 (7.5) | 42.3 (7.0)
  6 months | 42.0 (6.9) | 42.1 (7.2)
  Change at 6 months | -0.7 (8.6) | -0.2 (8.5)

6. Secondary Outcome: Change in Quality of Life as Assessed With the Short Form-12- Physical Component
Description: as for outcome 5
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 39.0 (8.2) | 40.1 (7.7)
  6 months | 40.4 (8.3) | 40.4 (7.9)
  Change at 6 months | 1.4 (7.7) | 0.3 (8.1)

7. Secondary Outcome: Change in Medication Use Self-efficacy Score as Measured by SEAMS Scale and the Perceived Diabetes Self-Management Scale, Which is Associated With A1c
Description: Medication use self-efficacy scores for range from 13-39; higher scores indicate higher levels of self-efficacy for medication adherence.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 31.9 (5.6) | 32.2 (6.0)
  6 months | 33.9 (5.1) | 33.1 (5.5)
  Change at 6 months | 2.0 (5.6) | 0.9 (5.0)

8. Secondary Outcome: Change in Diabetes-Specific Quality of Life
Description: Diabetes specific quality of life will be assessed using the validated Diabetes Distress Scale.The DDS is a 17-item instrument that measures diabetes-related emotional distress. Participants rate the degree to which each item is problematic for them on a 6-point Likert scale, from 1 (no problem) to 6 (serious problem). A score of 3 or greater = moderate distress.
Time Frame: Baseline, 6 months
Population: 39 participants in the peer coaching arm and 34 participants in the usual care arm were not analyzed because the participants were unable to be contacted, had health reasons, or did not have time.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 236
Scores on a scale
  Baseline | 2.6 (1.3) | 2.3 (1.3)
  6 months | 1.9 (1.1) | 2.0 (1.2)
  Change at 6 months | -0.6 (1.3) | -0.3 (1.3)

9. Secondary Outcome: Number of Physician Office Visits 6 Months
Time Frame: 6 months
Population: This data was not collected.
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Hospital Stays at 6 Months
Time Frame: 6 months
Population: This data was not collected.
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Emergency Visits at 6 Months
Time Frame: 6 months
Population: This data was not collected.
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Diabetes Medication Counts
Description: Change in number of diabetes medications.
Time Frame: Baseline, 6 months
Population: 44 participants in the peer coaching arm and 38 participants in the usual care arm were not analyzed because the participants were unable to be contacted, had health reasons, or did not have time.
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 159 | 232
Medications
  Baseline | 1.4 (0.7) | 1.3 (0.6)
  6 months | 1.3 (0.6) | 1.3 (0.6)
  Change at 6 months | -0.04 (0.5) | 0.004 (0.6)

13. Other Pre Specified Outcome: Change in Medication Beliefs- Harm (Beliefs That Medications Are Harmful)
Description: Beliefs about medications questionnaire scores range from 5-25; higher scores indicate stronger beliefs.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 10.6 (2.7) | 9.8 (2.8)
  Follow-up | 9.8 (2.7) | 9.7 (2.8)
  Change | -0.8 (2.5) | -0.1 (2.8)

14. Other Pre Specified Outcome: Change in Medication Beliefs- Overuse (Concerns About the Way Doctors Use Medications)
Description: Beliefs about medications questionnaire scores range from 5-25; higher scores indicate stronger beliefs.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 13.3 (3.2) | 12.7 (3.4)
  Follow-up | 12.6 (3.4) | 12.6 (3.4)
  Change | -0.6 (3.3) | -0.1 (3.3)

15. Other Pre Specified Outcome: Change in Medication Beliefs-Necessity (Beliefs About the Necessity of Medications)
Description: Beliefs about medications questionnaire scores range from 5-25; higher scores indicate stronger beliefs.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 19.1 (3.6) | 19.6 (3.9)
  Follow-up | 20.0 (3.9) | 19.4 (4.2)
  Change | 0.9 (3.5) | -0.2 (3.7)

16. Other Pre Specified Outcome: Change in Medication Beliefs- Concerns (Concerns About the Negative Effects of Medications)
Description: Beliefs about medications questionnaire scores range from 5-25; higher scores indicate stronger beliefs.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Peer Coaching | Usual Care
Number analyzed (Participants) | 164 | 239
Scores on a scale
  Baseline | 15.4 (3.9) | 14.9 (4.2)
  Follow-up | 14.0 (3.8) | 14.7 (8.9)
  Change | -1.5 (4.0) | -0.2 (3.9)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Peer Coaching | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/270
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/270
Other Adverse Events (participants affected / at risk) | 0/203 | 0/270

LIMITATIONS AND CAVEATS:
Delays in follow-up data collection for some participants could impact the A1c findings, medication adherence was not measured using objective means, and participants in this sample were mostly women, possibly limiting generalizability to men.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02274844/Prot_SAP_003.pdf